CLINICAL TRIAL: NCT02556359
Title: Consequences of DNA Repair and Telomere Defects on the Function of the Immune System: Application to CVID and Immune Deficiencies With Dysmorphic Syndromes
Acronym: IMMUNEREP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: RTC13005
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Immune Deficiency and Early BMF in Childhood
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained as a source of DNA and viable lymphocytes for functional studies. Blood will be sent to the laboratory of Dr JP de Villartay, INSERM UMR1163, Genome Dynamics in the Immune System, Université Paris Descartes - Sorbonne Paris Cité, Institut Imagine, 24 boulevard du Montparnasse, 75015 PARIS. Functional studies will be performed immediately.
  A portion of the blood sample taken as part of the research will be included in a biological collection: B-EBV cell lines will be derived from patients and their parents. EBV-B cell lines will be established by Centre de Ressource Biologique (CRB, Hôpital Necker - Enfants Malades, Bâtiment IMAGINE 1er étage, 149, rue de Sèvres - 75 743 PARIS CEDEX 15, under the supervision of Dr Marie-Alexandra Alyanakian & Anne Esling & Christine Gouarin). Skin biopsies will be obtained from patients to derive fibroblast lines at CRB.
Oversight: Data Monitoring Committee: No

SUMMARY:
The molecular mechanisms participating in the various aspects of the DNA Damage Response (DDR) are absolutely essential to maintain the genome dynamics essential to all living organisms. The most commonly studied consequence of faulty DDR is genome instability participating in cancer onset. In the present proposal, we wish to explore another aspect of DDR, not relevant to cancer, which is its absolute requirement at several key steps of the development, maturation, and function of the immune system.

The most "spectacular" consequences of faulty DNA repair processes with respect to the immuno-hematopoietic tissue are the complete block of B and T lymphocytes maturation owing to defective DNA joining phase during V(D)J recombination resulting in patients with Severe Combined Immune Deficiency (SCID).

The objectives of this study are to increase our knowledge on the role of the various DNA repair processes in the development, the maintenance, and the function of the immune system and thus, to better understand why and how dysfunctions of these DNA repair processes result in human severe conditions such as CVID, LOCID or other manifestations of immune disorders such as autoimmunity.

The explorations of DNA repair mechanisms in the patients will allow us to establish the genetic diagnosis in some patients with until now undefined molecular diagnosis. This is of immediate importance for the patients and their families, as it not only contributes to a better understanding of the patients' condition, but also allows providing genetic counseling for the families.

ELIGIBILITY:
Inclusion Criteria:

* Immune Deficiency and early BMF in childhood
* Common Variable Immunodeficiency (CVID)
* Genetic patients

Exclusion Criteria:

* Refusal to consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient presenting clinical immune deficiency and at least one associated feature hinting at a possible DNA repair defect, such as microcephaly, growth retardation starting in utero, distinctive facial appearance ("bird-like face"), developmental delay, cerebellar degeneration, UV light sensitivity, premature aging, dystrophic nails, dental abnormalities, hair anomalies, pancytopenia and/or bone marrow failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-07 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
DNA abnormailities | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, Paris, France